CLINICAL TRIAL: NCT04287582
Title: The Evaluation of Muscle Activation in Climbing up Stairs Activity in Children With Duchenne Muscular Dystrophy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Merve Bora, Principal Investigator, Hacettepe University
Other Study IDs: GO 19/323
Record Dates: First submitted 2020-02-23; First posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: duchenne muscular dystrophy; surface electromyography; muscle activation; stair climbing
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Level 1 DMD: According to Brooke Lower Extremity Functional Classification Level 1
  Interventions: Other: Electromyographic device
- Level 2-3 DMD: According to Brooke Lower Extremity Functional Classification Level 2 or 3
  Interventions: Other: Electromyographic device
- Healthy Group: healthy children with similar demographic characteristics with children with DMD
  Interventions: Other: Electromyographic device

INTERVENTIONS:
Other: Electromyographic device — An 8-channel surface EMG system (DELSYS Trigno Wireless System) will be used to measure signals from muscles during stair climbing activity by surface electromyography measurements.Surface EMG measurements will be carried out during stair climbing activity without any intervention in the body. Surface EMG electrodes will be placed bilaterally in the vastus lateralis, biceps femoris, tibialis anterior and gastrocnemius medialis muscles.

SUMMARY:
Children with Duchenne Muscular Dystrophy (DMD) have difficulties towards the end of the ambulatory period, especially in activities that require lower extremity proximal muscle strength such as walking, climbing stairs, standing up without sitting. Stair climbing / descending activity is a complex activity that requires joint stability, correct muscle synergy and timing. When the literature is examined; It has been observed that the performance of stair climb up and down activity in individuals with neuromuscular disease has been evaluated with various clinical applications. In recent studies, there are surface electromyography (EMG) studies evaluating various aspects of stair climbing and descending activity.

Surface EMG; is a technique for neuromuscular evaluations that is frequently used in both research and clinical applications, noninvasive, and can be used in areas such as neurophysiology, sports science and rehabilitation.

Our study was planned to examine the muscle activations in the lower limb muscles involved in climbing up stairs activity in children with DMD and to compare healthy children with children with DMD and children with different levels of DMD.

Hypothesis originating from the investigation:

H0: There is no difference in the muscle activations measured by surface electromyography (EMG) of the involved lower extremity muscles during climbing up stairs activity between level 1 and level 2-3 children with early DMD.

H1: There is a difference in the muscle activations measured by surface electromyography (EMG) of the involved lower extremity muscles during climbing up stairs activity between level 1 and level 2-3 children with early DMD.

H2: There is no difference in the muscle activations measured by surface electromyography (EMG) of the involved lower extremity muscles during climbing up stairs activity between children with DMD and healthy children.

H3: There is a difference in the muscle activations measured by surface electromyography (EMG) of the involved lower extremity muscles during climbing up stairs activity between children with DMD and healthy children.

DETAILED DESCRIPTION:
In our study, children will be assessed using the surface Electromyography (EMG) device by using electrodes placed in the relevant lower limb muscles that take part during the stair climbing activity.

The study included 10 children with DMD levels were 1 and 10 children with DMD levels were 2-3 according to the Brooke Lower Limb Functional Classification scale and 10 healthy children.

Muscle activation of vastus lateralis, biceps femoris, tibialis anterior and gastrocnemius medialis muscles will be measured by superficial electromyographic measurement. Muscle activation according to SENIAM (surface EMG for a non-invasive assessment of muscles) for will be evaluated.

Stair climbing activity will be performed 3 times and at 1 minute intervals.

ELIGIBILITY:
Inclusion Criteria:

Children with DMD:

* Having been diagnosed with Duchenne Muscular Dystrophy by a pediatric neurologist,
* Volunteering to participate in the study,
* Being in the 5-12 age range
* According to the Brooke Lower Limb Functional Classification developed for classifying lower extremity functions of children with DMD, it should be between level 1-3 (children who continue ambulation and can go up and down with assisted / unassisted stairs),
* To be able to cooperate with the instructions of the physiotherapist

Healthy Group:

* Not having a known acute or chronic illness
* The children with DMD included in the study have similar demographic characteristics (age, height, weight, body mass index),
* The physiotherapist should cooperate with the instructions.

Exclusion Criteria:

Children with DMD:

* Have undergone any lower limb injuries and / or surgery,
* Started steroid treatment in the last 6 months,
* Having any systemic disease other than DMD,
* Not having permission from his family and himself.

Healthy Group:

* Having had any injury and / or surgery ,
* Children with DMD have relatives,
* Not having permission from his family and himself

Ages: 5 Years to 12 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study included 20 children with DMD applied in the Hacettepe University Pediatric Neuromuscular Disorders Unit and 10 children aged 5-12 years living in Ankara who do not have any disease.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-04-03 (Actual); Primary Completion 2020-03-07 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Surface Electromyographic Measurement | 40 minutes
  Muscle Activation Measurement It is an 8-channel system for measuring signals come from muscles (Delsys)

SECONDARY OUTCOMES:
Muscle Strength Measurement | 15 minutes
  A quantitative and objective method for assessment of muscular strength using a portable hand held dynamometer. Muscle strength measurement included lower limb and trunk muscles.
Timed Performance Test | 20 minutes
  Timed function tests included time taken to stand from a supine position, time taken to walk 10 m, time taken to climb 4 standard-sized stairs and time taken to descend 4 standard-sized stairs.
Muscle shortness assessment | 10 minutes
  Shortening assessment of trunk and lower extremity muscles measurement included back extensors, hamstring, hip flexors, quadriceps and gastrocnemius muscles.
Six minute walk test | 6 minutes
  Children were asked to walk during 6 minutes as fast as possible at a 25 meter corridor.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Uchikawa K, Liu M, Hanayama K, Tsuji T, Fujiwara T, Chino N. Functional status and muscle strength in people with Duchenne muscular dystrophy living in the community. J Rehabil Med. 2004 May;36(3):124-9. doi: 10.1080/16501970410023461. PMID 15209455
- [Background] Bakker JP, De Groot IJ, Beelen A, Lankhorst GJ. Predictive factors of cessation of ambulation in patients with Duchenne muscular dystrophy. Am J Phys Med Rehabil. 2002 Dec;81(12):906-12. doi: 10.1097/00002060-200212000-00004. PMID 12447089
- [Background] Rainoldi A, Melchiorri G, Caruso I. A method for positioning electrodes during surface EMG recordings in lower limb muscles. J Neurosci Methods. 2004 Mar 15;134(1):37-43. doi: 10.1016/j.jneumeth.2003.10.014. PMID 15102501
- [Background] Ropars J, Lempereur M, Vuillerot C, Tiffreau V, Peudenier S, Cuisset JM, Pereon Y, Leboeuf F, Delporte L, Delpierre Y, Gross R, Brochard S. Muscle Activation during Gait in Children with Duchenne Muscular Dystrophy. PLoS One. 2016 Sep 13;11(9):e0161938. doi: 10.1371/journal.pone.0161938. eCollection 2016. PMID 27622734
- [Background] Hermens HJ, Freriks B, Disselhorst-Klug C, Rau G. Development of recommendations for SEMG sensors and sensor placement procedures. J Electromyogr Kinesiol. 2000 Oct;10(5):361-74. doi: 10.1016/s1050-6411(00)00027-4. PMID 11018445
- [Derived] Bora M, Yalcin A, Bulut N, Yilmaz O, Karaduman A, Topuz S, Alemdaroglu-Gurbuz I. Investigation of surface electromyography amplitude values during stair climbing task in children with Duchenne muscular dystrophy. Neurol Sci. 2022 Apr;43(4):2791-2801. doi: 10.1007/s10072-021-05643-y. Epub 2021 Oct 4. PMID 34608577
- See also: SENIAM — http://www.seniam.org/